CLINICAL TRIAL: NCT01808313
Title: An Open Label Phase IIIb Study to Evaluate Efficacy and Safety of Ambrisentan in Chinese Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Efficacy Study of Ambrisentan in Chinese Patients With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115812
Record Dates: First submitted 2013-02-28; First posted 2013-03-11 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Vascular Disease
MeSH Terms: conditions — Vascular Diseases | interventions — ambrisentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ambrisentan (Experimental): ambrisentan 5 mg will be administered to eligible subjects for 12 weeks
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — Ambrisentan 5 mg will be administered to eligible subjects for 12 weeks

SUMMARY:
This open label, single-arm, non-controlled, multicentre study will determine the effect of ambrisentan on exercise capacity (6MWT) in Chinese subjects with PAH. The study consists of a screening period of 4 weeks, a 12-week primary evaluation period (PEP) and a 12-week dose-adjustment period (DAP). Ambrisentan 5 mg will be administered to eligible subjects for 12 weeks (PEP).

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) consists of a group of progressive and incurable diseases of the pulmonary vasculature. These are characterised by profound vasoconstriction and abnormal proliferation of smooth muscle cells in the walls of the pulmonary arteries, which leads to a progressive increase in pulmonary vascular resistance (PVR) and sustained elevations in pulmonary artery pressure (PAP). A variety of drug classes have been used to treat PAH but no single compound has yet been shown to be effective in treating all patients with the disease. Three widely used treatment options are calcium channel blockers (CCBs), diuretics and anticoagulants but all have varying responses.There is a lack of clinical data on ambrisentan among the Chinese population,Ambrisentan is conditionally approved for the treatment of PAH in China.A clinical trial with a minimum of 100 patients in the ambrisentan arm was requested by SFDA.Several PAH medications have been approved in China, so a placebo-controlled study is not ethically appropriate while an active control non-inferiority design is unfeasible due to sample size requirements and inconsistency in indications.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning study-related procedures.
* Subject must be between 18-75 years of age, inclusive, at the Screening Visit.
* Subjects must weight ≥40 kg at the Screening Visit.
* Subjects must have symptomatic or severe PAH (WHO functional class II or III) and be categorised as class 1 PAH (defined by the Updated Clinical Classification of Pulmonary Hypertension 2009), due to iPAH, congenital heart disease-congenital heart defects repaired greater than 1 year prior to screening (i.e., atrial septal defects, ventricular septal defects or patent ductus arteriosus) or CTD-related PAH (e.g., limited scleroderma, diffuse scleroderma, mixed CTD, systemic lupus erythematosus or overlap syndrome).

NOTE: subjects with portopulmonary hypertension and pulmonary venoocclusive disease are NOT eligible for the study.

* Subjects must have had a right heart catheterisation within 6 months prior to screening and meet all of the following haemodynamic criteria:

  1. Mean PAP ≥ 25 mmHg.
  2. A PVR ≥ 240 dyn/sec/cm5.
  3. A PCWP or left ventricular (LV) end-diastolic pressure of ≤ 15 mmHg.
* Subjects must be able to walk a distance of at least 150 m but no more than 450 m. In addition, the screening and baseline 6MWT test values must not vary by greater than 10% (calculated using (baseline - screening)/screening with the result to be between -0.1 and 0.1).
* Subjects must meet both of the following pulmonary function criteria. The tests should have been completed no more than 24 weeks prior to the Screening Visit, if not performed within the previous 24 weeks, the test must be completed at Day 0:

  1. Total lung capacity (TLC) ≥ 60% of predicted normal.
  2. Forced expiratory volume in one second (FEV1) ≥ 55% of predicted normal.
* Subjects receiving CCBs must be on stable therapy (i.e., the dose level does not need to change to maintain disease control) for at least 1 month prior to the Screening Visit.
* Subjects receiving 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (i.e., statins) must be on stable therapy (i.e., the dose level does not need to change to maintain disease control) for at least 12 weeks prior to the Screening Visit.
* Female subjects of childbearing potential must have a negative pregnancy test at the Screening Visit and Day 0.
* Female subjects of childbearing potential who are sexually active must agree to use two reliable methods of contraception (as described in Appendix 3 ) from the Screening Visit until study completion and for at least 30 days following the last dose of IP. Subjects who have had a Copper T 380A intrauterine device (IUD) or LNg 20 IUD inserted are not required to use an additional method of contraception.
* Subject must agree not to participate in a clinical study involving another IP or device throughout this study.

Exclusion Criteria:

* The subject has received PAH therapy (PDE-5 inhibitors, ERA, chronic prostanoid*) within 4 weeks prior to the Screening Visit.

  *Prostanoid use is classed as chronic when treatment continues for more than 7 days.
* The subject has received intravenous inotropes (e.g., dopamine, dobutamine) within 2 weeks prior to the Screening Visit.
* The subject has previously been discontinued from ERA treatment (e.g., bosentan) due to safety or tolerance issues other than those associated with liver function abnormalities.
* The subject has a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value that is >2 x the upper limit of normal (ULN) at the Screening Visit.
* The subject has serum bilirubin value that is >1.5 x ULN at the Screening Visit.
* The subject has severe hepatic impairment (Child-Pugh class C with or without cirrhosis) at the Screening Visit.
* The subject has severe renal impairment (creatinine clearance <30 mL/min) at the Screening Visit.
* The subject has clinically significant anaemia, defined as haemoglobin concentration <10 g/dL or haematocrit <30% at the Screening Visit.
* The subject has a laboratory result, physical examination finding, medical history incident or other finding, which is a contraindication for treatment with an ERA. Contraindications for treatment include, but are not limited to, evidence of elevated liver functions test or previously experiencing an event that would be defined as a serious AE (SAE) in a clinical trial (see Section 6.3.3.2), which was attributed to treatment with an ERA.
* The subject has severe hypotension (either diastolic blood pressure <50 mmHg or systolic blood pressure <90 mmHg).
* The subject has, in the opinion of the Investigator, clinically significant aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, life-threatening cardiac arrhythmias, significant LV dysfunction (defined as LV ejection fraction <45%), LV outflow obstruction, symptomatic coronary artery disease, autonomic hypotension or fluid depletion.
* The subject has a history of malignancies within the past 5 years, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* The subject has cardiovascular, liver, renal, haematological, gastrointestinal, immunological, endocrine, metabolic or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject.
* A female subject who is pregnant or breastfeeding.
* The subject has demonstrated non-compliance with previous medical regimens or is unable to comply with the procedures described in this protocol.
* The subject has a history of abusing alcohol or drugs of abuse (including amphetamines, methamphetamines, opiates, cannabinoids, cocaine, benzodiazepines or barbiturates) within 12 months prior to the Screening Visit. Use of such drugs if prescribed by a Doctor and used according to the prescription would not exclude a subject.
* The subject has participated in a clinical study involving another IP or device within 4 weeks or five half-lives of an IP, whichever is longer, before the Screening Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2014-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- China (8):
  - GSK Investigational Site, Harbin, Heilongjiang
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Hunan, Hunan
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai

REFERENCES:
- [Derived] Zhao QH, Peng FH, Yu ZX, Zhang GC, Ji QS, Wang Y, Liu JM, Huo Y, Zeng XF, Li JH, Zi L, Jing ZC. Effect of ambrisentan on echocardiographic and Doppler measures from patients in China with pulmonary arterial hypertension. Expert Rev Cardiovasc Ther. 2020 Sep;18(9):643-649. doi: 10.1080/14779072.2020.1807942. Epub 2020 Sep 29. PMID 32799568
- [Derived] Li M, Jing ZC, Li Y, Huo Y, Yu Z, Zhang G, Zhu P, Liu J, Ji Q, Wu B, Zhong J, Wang P, Zhu W, Zeng X. Efficacy and safety of ambrisentan in Chinese patients with connective tissue disease-pulmonary arterial hypertension: a post-hoc analysis. BMC Cardiovasc Disord. 2020 Jul 17;20(1):339. doi: 10.1186/s12872-020-01591-1. PMID 32680480
- [Derived] Huo Y, Jing ZC, Zeng XF, Liu JM, Yu ZX, Zhang GC, Li Y, Wang Y, Ji QS, Zhu P, Wu BX, Zheng Y, Wang PP, Li J. Evaluation of efficacy, safety and tolerability of Ambrisentan in Chinese adults with pulmonary arterial hypertension: a prospective open label cohort study. BMC Cardiovasc Disord. 2016 Oct 22;16(1):201. doi: 10.1186/s12872-016-0361-9. PMID 27770771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 134 participants were enrolled and received at least one dose of study medication. 133 participants comprised the Intent-to-Treat (ITT) Population (all participants that received at least one dose of study treatment and had an efficacy assessment performed both at Baseline and after administration of the study treatment).
Groups:
- Ambrisentan: Participants received one tablet of 5 milligrams (mg) ambrisentan (AMB) once daily (QD) for the first 12 Weeks. After 12 Weeks, the AMB dose was titrated to either one tablet of 5 mg QD or one tablet of 10 mg QD, as determined by the investigator for another 12 Weeks.
Period: Overall Study
Arm/Group | Ambrisentan
Started | 133
Completed | 123
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 2
Not completed — Met Protocol-defined Stopping Criteria | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 20
Race/Ethnicity, Customized [Number; unit: Particiopants]
  Asian-East Asian Heritage | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6-minutes Walk Test (6MWT) at Week 12
Description: The 6MWT measures the distance that a participant can walk in a period of 6 minutes. Change from Baseline was calculated as the Week 12 value minus the Baseline value. Baseline 6MWT comprised of an average of the last two consecutive measurements prior to dosing that varied by not greater than 10 percent (%). If only one measurement was available, that measurement was used as the Baseline value. The last observation carried forward method was used to impute missing values.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication and had an efficacy assessment performed both at Baseline and after administration of the study medication
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Meters | 53.59 (64.494)
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 53.59, 95% CI 2-sided [42.53 to 64.66]

2. Secondary Outcome: Change From Baseline in 6MWT at Week 24
Description: The 6MWT measures the distance that a participant can walk in a period of 6 minutes. Change from Baseline was calculated as the Week 24 value minus the Baseline value. Baseline 6MWT comprised of an average of the last two consecutive measurements prior to dosing that varied by not greater than 10%. If only one measurement was available, that measurement was used as the Baseline value. The last observation carried forward method was used to impute missing values.
Time Frame: Baseline and Week 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Meters | 64.36 (91.173)
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 64.36, 95% CI 2-sided [48.72 to 80.00]

3. Secondary Outcome: Number of Participants With a Change From Baseline in Their World Health Organization (WHO) Functional Classification (FC) at Weeks 12 and 24
Description: The WHO FC was determined by the investigator as follows: Class I- Participants with pulmonary hypertension (PH) but without resulting limitation of physical activity, II- Participants with PH resulting in slight limitation of physical activity, III- Participants with PH resulting in marked limitation of physical activity, IV- Participants with PH with inability to carry out any physical activity without symptoms. Changes from Baseline in functional class were summarized at Weeks 12 and 24. The number of participants improving by 2 classes, improving by 1 class, not changing, worsening by 1 class or worsening by 2 classes from Baseline at Weeks 12 and 24 were evaluated. The Baseline value was the last non-missing assessment value before treatment. Only participants with non-missing Baseline values and at least one non-missing post-Baseline value of the response variable were included. The last observation carried forward method was used to impute missing values.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Participants
  Improved by 2 classes at Week 12 | 0
  Improved by 1 class at Week 12 | 44
  Not changing at Week 12 | 84
  Worsened by 1 class at Week 12 | 4
  Worsened by 2 classes at Week 12 | 1
  Improved by 2 classes at Week 24 | 0
  Improved by 1 class at Week 24 | 51
  Not changing at Week 24 | 77
  Worsened by 1 class at Week 24 | 3
  Worsened by 2 classes at Week 24 | 2

4. Secondary Outcome: Change From Baseline in the Borg Dyspnea Index (BDI) at Weeks 12 and 24
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum). Change from Baseline was calculated as the Week 12 and 24 values minus the Baseline values. The BDI indicates the degree of exertion, breathlessness, fatigue, or difficulty breathing after completion of the 6MWT. The lower values, 0 as the lowest, indicates no exertion, fatigue, or breathlessness felt, and 10 would be the maximum amount of exertion felt as assessed by each participant. The last observation carried forward method was used to impute missing values.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
scores on a scale
  Week 12 | -0.34 (1.521)
  Week 24 | -0.22 (1.952)
Statistical Analysis 1: Comparison: Ambrisentan; Week 12; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Ambrisentan; Week 24; Test type: Superiority or Other; p = 0.003, Wilcoxon signed-rank test

5. Secondary Outcome: Change From Baseline in the N-Terminal Pro-B-Type Natriuretic Peptide at Weeks 12 and 24
Description: N-Terminal Pro-B-Type Natriuretic Peptide (NT-proBNP) is a surrogate maker of heart failure and was measured by a central laboratory. Mean change from Baseline at Weeks 12 and 24 were calculated as the Weeks 12 and 24 values minus the Baseline values.Observed data was analyzed (no imputation technique was performed for missing data). Log transformed mean change from Baseline at Weeks 12 and 24 data are summarized.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by number of participants [n]=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflect everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: log(ng/L)
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
log(ng/L)
  Week 12, n=123 | 0.44 (2.687)
  Week 24, n=122 | 0.37 (3.103)
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean Difference (Net) = 0.44, 95% CI 2-sided [0.366 to 0.519] — Week 12
Statistical Analysis 2: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [0.303 to 0.453] — Week 24

6. Secondary Outcome: Number of Participants With the Indicated Event, as an Assessment of Time to Clinical Worsening of Pulmonary Arterial Hypertension (PAH) up to Week 24, Assessed as the First Occurrence of a Particular Event
Description: Time to clinical worsening is defined as the time from Baseline to the first occurrence of death, lung transplantation, hospitalization for PAH treatment, atrial septostomy, or Investigational product (IP) discontinuation (discon) due to change to other PAH treatment. Time to clinical worsening was measured as the number of participants who experienced these events during 12 and 24 Weeks.
Time Frame: Baseline up to Week 24
Population: Safety Population: This population comprised of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Participants
  Death at Week 12 | 2
  Lung Transplant at Week 12 | 0
  Hospitalization for PAH at Week 12 | 0
  Atrial Septostomy at Week 12 | 0
  IP discon (additional medication) at Week 12 | 0
  Death at Week 24 | 3
  Lung Transplant at Week 24 | 0
  Hospitalization for PAH at Week 24 | 1
  Atrial Septostomy at Week 24 | 0
  IP discon (additional medication) at Week 24 | 0

7. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events and Adverse Events Leading to Discontinuation
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect, or important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: From the start of study treatment up to Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Participants
  Any AEs | 91
  Any SAEs | 11
  AEs leading to discontinuation | 4

8. Secondary Outcome: Number of Participants With Physical Examination Findings
Description: Complete physical examinations of each participant by the investigator were performed at the Screening Visit, Week 12 and Week 24 Visit/Early withdrawal visits. The physical examination included an examination of the following: general appearance, skin, head, ears, eyes, nose, throat, neck, thyroid, lymph nodes, cardiovascular system, respiratory system, abdomen, musculoskeletal system, neurological system and height. Physical examination summary results were not collected therefore there is no data to present for this outcome measure.
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Participants | NA — Summary data was not compiled for this outcome measure therefore there is no data to present.

9. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Heart Rate Values at Weeks 12 and 24
Description: Heart rate was measured in order to monitor vital signs by the 12-lead ECG at Baseline, Weeks 12 and 24. Change from Baseline in ECG heart rate is summarized for each post-Baseline assessment at Weeks 12 and 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last non-missing observed value before treatment.
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Ambrisentan
Number analyzed (Participants) | 128
Beats per minute
  Week 12, n=124 | -2.0 (16.65)
  Week 24, n=118 | -4.6 (14.68)

10. Secondary Outcome: Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval, QT Interval Corrected Bazett's Formula (QTcB) Values at Weeks 12 and 24
Description: The ECG parameters, PR interval, QRS duration, uncorrected QT interval, QTcB were measured at Baseline, Weeks 12 and 24. Change from Baseline in ECG heart rate is summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last non-missing observed value before treatment.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Milliseconds
  PR interval, Week 12, n=122 | 0.7 (16.55)
  PR interval, Week 24, n=117 | 1.5 (14.84)
  QRS duration, Week 12, n=124 | -1.5 (15.84)
  QRS duration, Week 24, n=118 | 0.7 (14.40)
  Uncorrected QT Interval, Week 12, n=124 | -0.7 (37.44)
  Uncorrected QT Interval, Week 24, n=118 | 6.8 (40.41)
  Corrected QTcB interval, Week 12, n=123 | -4.9 (29.74)
  Corrected QTcB interval, Week 24, n=117 | -1.5 (37.25)

11. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at the Indicated Time Points up to Week 24
Description: Blood pressure measurements (pre-6MWT and post-6MWT) were taken to monitor vital signs and included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at the Baseline, Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in SBP and DBP were summarized for each post-Baseline assessment upto Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last non-missing observed value before treatment.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Millimeters of mercury (mmHg)
  SBP; pre-6MWT; Week 4; n=131 | -1.6 (11.57)
  SBP; post-6MWT; Week 4; n=131 | 0.7 (15.36)
  SBP; pre-6MWT; Week 8; n=126 | -2.2 (13.89)
  SBP; post-6MWT, Week 8; n=126 | 2.3 (17.36)
  SBP; pre-6MWT; Week 12; n=126 | -1.9 (15.08)
  SBP; post-6MWT; Week 12; n=125 | 0.3 (18.23)
  SBP; pre-6MWT; Week 16; n=124 | -1.8 (14.55)
  SBP; post-6MWT; Week 16; n=123 | 1.7 (17.71)
  SBP; pre-6MWT; Week 20; n=122 | -3.3 (14.42)
  SBP; post-6MWT, Week 20; n=122 | 1.3 (18.07)
  SBP; pre-6MWT; Week 24; n=123 | -3.4 (15.14)
  SBP; post-6MWT; Week 24; n=123 | 1.0 (19.01)
  DBP; pre-6MWT; Week 4; n=131 | -3.2 (9.30)
  DBP; post-6MWT; Week 4; n=131 | -1.6 (11.19)
  DBP; pre-6MWT; Week 8; n=126 | -3.6 (9.73)
  DBP; post-6MWT; Week 8; n=126 | -1.8 (11.48)
  DBP; pre-6MWT; Week 12; n=126 | -3.5 (10.39)
  DBP; post-6MWT; Week 12; n=125 | -4.2 (12.84)
  DBP; pre-6MWT; Week 16; n=124 | -5.0 (11.66)
  DBP; post-6MWT; Week 16; n=123 | -3.0 (14.20)
  DBP; pre-6MWT; Week 20; n=122 | -4.6 (10.97)
  DBP; post-6MWT; Week 20; n=122 | -2.5 (14.37)
  DBP; pre-6MWT; Week 24; n=123 | -4.6 (12.35)
  DBP; post-6MWT; Week 24; n=123 | -2.5 (13.30)

12. Secondary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points up to Week 24
Description: Vital sign monitoring included heart rate measurements at (pre-6MWT and post-6MWT at the Baseline visit, Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in heart rate was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last non-missing value observed before treatment. At Baseline, Weeks 12 and 28, heart rate was recorded at the end of the 6MWT and at 1 minute (M), 2 M and 3 M, after completion of the 6MWT with the participants seated, and the time that heart rate recovered to the level of pre-6MWT.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Ambrisentan
Number analyzed (Participants) | 133
Beats per minute
  Heart Rate; pre-6MWT; Week 4; n=131 | -0.7 (12.12)
  Heart Rate; post-6MWT; Week 4; n=131 | -2.1 (18.26)
  Heart Rate; pre-6MWT; Week 8; n=126 | -1.2 (13.10)
  Heart Rate; post-6MWT, Week 8; n=126 | -0.2 (17.39)
  Heart Rate; pre-6MWT; Week 12; n=126 | -1.7 (12.27)
  Heart Rate; post-6MWT; Week 12; n=124 | 0.6 (18.23)
  Heart Rate; post-6MWT 1M; Week 12; n=124 | -0.9 (15.11)
  Heart Rate; post-6MWT 2 M; Week 12; n=124 | -2.2 (13.51)
  Heart Rate; post-6MWT 3 M; Week 12; n=125 | -1.2 (13.90)
  Heart Rate; Recovery to Pre-6MWT; Week 12; n=125 | -1.5 (12.50)
  Heart Rate; pre-6MWT; Week 16; n=124 | -2.6 (13.10)
  Heart Rate; post-6MWT; Week 16; n=123 | 0.5 (19.81)
  Heart Rate; pre-6MWT; Week 20; n=122 | -3.6 (12.45)
  Heart Rate; post-6MWT, Week 20; n=122 | 0.4 (20.82)
  Heart Rate; pre-6MWT; Week 24; n=123 | -0.8 (13.34)
  Heart Rate; post-6MWT; Week 24; n=123 | 3.4 (21.88)
  Heart Rate; post-6MWT 1 M; Week 24; n=121 | 0.3 (16.57)
  Heart Rate; post-6MWT 2 M; Week 24; n=121 | -0.5 (13.95)
  Heart Rate; post-6MWT 3 M; Week 24; n=122 | -0.2 (13.41)
  Heart Rate; Recovery to Pre-6MWT; Week 24; n=123 | -0.4 (13.39)

13. Secondary Outcome: Oral Temperature
Description: Oral temperature was used to monitor vital signs and collected at the Screening visit.
Time Frame: Baseline
Population: Safety Population
Measure: Mean (Full Range); unit: Celsius
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Celsius | 36.4 [35 to 37.3]

14. Secondary Outcome: Number of Participants With Shift From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST) and Total Bilirubin (BILT) up to Week 24
Description: Blood samples were collected for the measurement of ALT, ALP, AST and BILT at the Baseline visit and up to Week 24. Shift from Baseline (BL) was calculated as the individual maximum of post-BL value minus the BL value. The BL value is defined as the last pre-treatment value observed. Threshold values for the liver function test results, which were considered as potential values of clinical concern, were 3 times the upper limit of normal (ULN) for ALT, AST and ALP and 2 times the ULN for BILT. Maximum liver function abnormal values of post-BL are summarized.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Participants
  ALT; BL <=1 x ULN shift to >3 x ULN post-BL;n=133 | 0
  ALT; >1 x - <3 x ULN shift to >3 x ULN; n=133 | 3
  ALP; <=1 x ULN shift to >3 x ULN; n=132 | 0
  ALP; >1 x - <3 x ULN shift to >3 x ULN; n=132 | 0
  AST; <=1 x ULN shift to >3 x ULN; n=133 | 0
  AST; >1 x - <3 x ULN shift to >3 x ULN; n=133 | 2
  BILT; >1 x - <2 x ULN shift to >2 x ULN; n=133 | 1
  BILT; >1 x - <3 x ULN shift to >2 x ULN; n=133 | 3
  BILT; >1 x - >2 x ULN shift to >2 x ULN; n=133 | 1

15. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell (WBC) Count at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and WBC count at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and WBC count values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Giga cells per liter
  Basophils; Week 4; n=133 | -0.010 (0.0434)
  Basophils; Week 8; n=125 | -0.007 (0.0479)
  Basophils; Week12; n=125 | -0.009 (0.0438)
  Basophils; Week 16; n=125 | -0.006 (0.0484)
  Basophils; Week 20; n=125 | -0.002 (0.0366)
  Basophils; Week 24; n=123 | -0.002 (0.0792)
  Eosinophils; Week 4; n=133 | -0.0077 (0.0515)
  Eosinophils; Week 8; n=125 | -0.0004 (0.0588)
  Eosinophils; Week 12; n=125 | 0.0012 (0.0603)
  Eosinophils; Week 16; n=125 | 0.0126 (0.1466)
  Eosinophils; Week 20; n=125 | 0.0014 (0.0582)
  Eosinophils; Week 24; n=123 | 0.0014 (0.0854)
  Lymphocytes; Week 4; n=133 | -0.257 (0.5558)
  Lymphocytes; Week 8; n=125 | -0.201 (0.6116)
  Lymphocytes; Week 12; n=125 | -0.284 (0.5743)
  Lymphocytes; Week 16; n=125 | -0.295 (0.5821)
  Lymphocytes; Week 20; n=125 | -0.378 (0.6600)
  Lymphocytes; Week 24; n=123 | -0.363 (0.6897)
  Monocytes; Week 4; n=133 | -0.011 (0.1684)
  Monocytes; Week 8; n=125 | -0.013 (0.1713)
  Monocytes; Week 12; n=125 | -0.032 (0.1659)
  Monocytes; Week 16; n=125 | -0.019 (0.1665)
  Monocytes; Week 20; n=125 | -0.044 (0.1574)
  Monocytes; Week 24; n=123 | -0.000 (0.4885)
  Total Neutrophils; Week 4; n=133 | -0.4093 (1.7597)
  Total Neutrophils; Week 8; n=125 | -0.4209 (1.8660)
  Total Neutrophils; Week 12; n=125 | -0.5958 (1.8947)
  Total Neutrophils; Week 16; n=125 | -0.7201 (2.1282)
  Total Neutrophils; Week 20; n=125 | -0.9510 (2.0706)
  Total Neutrophils; Week 24; n=123 | -0.9247 (2.2646)
  Platelet Count; Week 4; n=133 | -4.80 (41.562)
  Platelet Count; Week 8; n=125 | -3.00 (49.357)
  Platelet Count; Week 12; n=125 | -1.56 (54.690)
  Platelet Count; Week 16; n=125 | -6.04 (50.227)
  Platelet Count; Week 20; n=125 | -7.89 (52.007)
  Platelet Count; Week 24; n=123 | -4.75 (45.181)
  WBC Count; Week 4; n=133 | -0.689 (1.9433)
  WBC count; Week 8; n=125 | -0.642 (2.1480)
  WBC count; Week 12; n=125 | -0.925 (2.1708)
  WBC Count; Week 16; n=125 | -1.050 (2.3951)
  WBC count; Week 20; n=125 | -1.387 (2.2706)
  WBC count; Week 24; n=123 | -1.342 (2.5167)

16. Secondary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of hemoglobin at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the hemoglobin count values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Grams per liter
  Hemoglobin; Week 4; n=133 | -7.46 (11.345)
  Hemoglobin; Week 8; n=125 | -6.80 (13.642)
  Hemoglobin; Week12; n=125 | -6.29 (14.269)
  Hemoglobin; Week 16; n=125 | -6.87 (14.245)
  Hemoglobin; Week 20; n=125 | -8.19 (14.862)
  Hemoglobin; Week 24; n=123 | -6.56 (14.724)

17. Secondary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of hematocrit at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the hematocrit values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is defined as the last Pre-treatment value observed. The unit of measure is defined as the proprtion of red blood cells in blood.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Proportion of 1
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Proportion of 1
  Hematocrit; Week 4; n=133 | -0.0168 (0.0587)
  Hematocrit; Week 8; n=125 | -0.0209 (0.0412)
  Hematocrit; Week12; n=125 | -0.0180 (0.0420)
  Hematocrit; Week 16; n=125 | -0.0179 (0.0443)
  Hematocrit; Week 20; n=125 | -0.0220 (0.0459)
  Hematocrit; Week 24; n=123 | -0.0176 (0.0422)

18. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of mean corpuscle hemoglobin at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the hemoglobin values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Picogram
  Mean Corpuscle Hemoglobin; Week 4; n=133 | 0.258 (1.4064)
  Mean Corpuscle Hemoglobin; Week 8; n=125 | 0.405 (1.5405)
  Mean Corpuscle Hemoglobin; Week12; n=125 | 0.347 (2.1082)
  Mean Corpuscle Hemoglobin; Week 16; n=125 | 0.185 (2.0053)
  Mean Corpuscle Hemoglobin; Week 20; n=125 | 0.019 (2.0040)
  Mean Corpuscle Hemoglobin; Week 24; n=123 | -0.035 (2.0831)

19. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of mean corpuscle volume at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the mean corpuscle volume values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Femtoliters
  Mean corpuscle volume; Week 4; n=133 | 0.906 (2.8849)
  Mean corpuscle volume; Week 8; n=125 | 1.362 (3.8958)
  Mean corpuscle volume; Week12; n=125 | 0.485 (7.4220)
  Mean corpuscle volume; Week 16; n=125 | 0.725 (6.6333)
  Mean corpuscle volume; Week 20; n=125 | 0.587 (4.7209)
  Mean corpuscle volume; Week 24; n=123 | 0.392 (4.8609)

20. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of RBC count at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the red blood cell count values were summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Trillion cells per liter
  RBC count; Week 4; n=133 | -0.2773 (0.3678)
  RBC count; Week 8; n=125 | -0.2987 (0.4781)
  RBC count; Week12; n=125 | -0.2520 (0.4672)
  RBC count; Week 16; n=125 | -0.2595 (0.5066)
  RBC count; Week 20; n=125 | -0.2733 (0.5414)
  RBC count; Week 24; n=123 | -0.2182 (0.4802)

21. Secondary Outcome: Change From Baseline in Albumin, Globulin and Total Protein at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of albumin, globulin and total protein at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the albumin, globulin and total protein values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Grams per liter
  Albumin; Week 4; n=132 | 1.01 (4.274)
  Albumin; Week 8; n=126 | 1.09 (3.717)
  Albumin; Week12; n=126 | 1.09 (4.105)
  Albumin; Week 16; n=126 | 1.05 (4.098)
  Albumin; Week 20; n=121 | 0.64 (4.625)
  Albumin; Week 24; n=120 | 1.31 (4.390)
  Globulin; Week 4; n=112 | -1.63 (5.083)
  Globulin; Week 8; n=106 | -2.17 (6.083)
  Globulin; Week12; n=107 | -2.38 (6.456)
  Globulin; Week 16; n=107 | -2.24 (6.120)
  Globulin; Week 20; n=103 | -2.57 (6.126)
  Globulin; Week 24; n=103 | -2.25 (6.251)
  Total Protein; Week 4; n=132 | -1.19 (9.058)
  Total Protein; Week 8; n=127 | -1.25 (8.555)
  Total Protein; Week12; n=126 | -1.57 (8.835)
  Total Protein; Week 16; n=126 | -1.37 (7.854)
  Total Protein; Week 20; n=122 | -2.60 (10.129)
  Total Protein; Week 24; n=121 | -0.91 (8.841)

22. Secondary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), creatine kinase (CK), gamma glutamyl transferase (GGT) and lactate dehydrogenase (LDH) at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the ALP, ALT, AST, CK, GGT and LDH values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
International units per liter
  ALP; Week 4; n=131 | -4.20 (14.945)
  ALP; Week 8; n=124 | -6.19 (16.612)
  ALP; Week12; n=125 | -6.79 (16.815)
  ALP; Week 16; n=122 | -4.47 (18.916)
  ALP; Week 20; n=124 | -5.99 (18.255)
  ALP; Week 24; n=121 | -2.95 (23.104)
  ALT; Week 4; n=133 | 0.07 (20.479)
  ALT; Week 8; n=127 | -1.58 (20.411)
  ALT; Week12; n=127 | -5.69 (16.770)
  ALT; Week 16; n=126 | -5.33 (16.064)
  ALT; Week 20; n=125 | -5.44 (19.143)
  ALT; Week 24; n=123 | -5.62 (15.734)
  AST; Week 4; n=132 | 0.18 (24.671)
  AST; Week 8; n=127 | -1.55 (13.848)
  AST; Week12; n=127 | -3.51 (13.835)
  AST; Week 16; n=125 | -4.03 (12.710)
  AST; Week 20; n=125 | -3.80 (15.021)
  AST; Week 24; n=123 | -3.63 (12.091)
  CK; Week 4; n=129 | -1.78 (35.099)
  CK; Week 8; n=123 | 11.21 (182.414)
  CK; Week12; n=124 | 1.62 (105.342)
  CK; Week 16; n=121 | 0.07 (100.783)
  CK; Week 20; n=120 | -1.79 (86.528)
  CK; Week 24; n=116 | 0.32 (89.377)
  GGT; Week 4; n=131 | -4.67 (46.013)
  GGT; Week 8; n=127 | -10.91 (49.174)
  GGT; Week12; n=127 | -15.82 (52.509)
  GGT; Week 16; n=124 | -13.98 (55.130)
  GGT; Week 20; n=125 | -20.42 (58.287)
  GGT; Week 24; n=122 | -21.84 (56.557)
  LDH; Week 4; n=122 | -20.45 (53.720)
  LDH; Week 8; n=118 | -19.24 (80.068)
  LDH; Week12; n=118 | -28.15 (77.867)
  LDH; Week 16; n=117 | -29.37 (82.565)
  LDH; Week 20; n=117 | -26.65 (81.007)
  LDH; Week 24; n=113 | -27.38 (74.551)

23. Secondary Outcome: Mean Change From Baseline in Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of direct bilirubin, total bilirubin, creatinine and uric acid at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the direct bilirubin, total bilirubin, creatinine and uric acid values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Micromoles per liter
  Direct Bilirubin; Week 4; n=131 | -0.326 (2.0821)
  Direct Bilirubin; Week 8; n=126 | -0.538 (2.5429)
  Direct Bilirubin; Week12; n=127 | -0.787 (2.5038)
  Direct Bilirubin; Week 16; n=126 | -0.778 (2.7692)
  Direct Bilirubin; Week 20; n=125 | -0.780 (2.5072)
  Direct Bilirubin; Week 24; n=122 | -0.752 (2.7299)
  Total Bilirubin; Week 4; n=131 | -0.72 (5.903)
  Total Bilirubin; Week 8; n=127 | -1.12 (6.089)
  Total Bilirubin; Week12; n=127 | -0.49 (17.178)
  Total Bilirubin; Week 16; n=126 | -1.49 (6.866)
  Total Bilirubin; Week 20; n=125 | -1.65 (6.329)
  Total Bilirubin; Week 24; n=123 | -1.25 (6.927)
  Creatinine; Week 4; n=133 | -1.924 (10.1256)
  Creatinine; Week 8; n=127 | -1.968 (10.7823)
  Creatinine; Week12; n=127 | -0.759 (9.2949)
  Creatinine; Week 16; n=126 | -0.847 (10.0814)
  Creatinine; Week 20; n=125 | -0.970 (9.3502)
  Creatinine; Week 24; n=123 | -0.217 (9.9447)
  Uric Acid; Week 4; n=129 | -13.289 (82.7246)
  Uric Acid; Week 8; n=125 | -13.159 (87.0456)
  Uric Acid; Week12; n=125 | -16.580 (83.7145)
  Uric Acid; Week 16; n=124 | -16.149 (87.9857)
  Uric Acid; Week 20; n=119 | -24.584 (94.9378)
  Uric Acid; Week 24; n=121 | -13.168 (95.0694)

24. Secondary Outcome: Change From Baseline in Calcium, Cholesterol, Chloride, Glucose, Potassium, Magnesium, Sodium, Inorganic Phosphorus, Triglycerides and Urea/Blood Urea Nitrogen (BUN) at the Indicated Time Points up to Week 24
Description: Blood samples were collected for the measurement of calcium, cholesterol, chloride, glucose, potassium, magnesium, sodium, inorganic phosphorus, triglycerides and urea/Bun at the Baseline visit and Weeks 4, 8, 12, 16, 20 and 24. Change from Baseline in the calcium, cholesterol, chloride, glucose, potassium, magnesium, sodium, inorganic phosphorus, triglycerides and urea/BUN values were summarized for each post-Baseline assessment until Week 24. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Millimoles per liter
  Calcium; Week 4; n=132 | -0.009 (0.1321)
  Calcium; Week 8; n=127 | -0.020 (0.1386)
  Calcium; Week12; n=127 | -0.008 (0.1340)
  Calcium; Week 16; n=126 | -0.015 (0.1470)
  Calcium; Week 20; n=124 | -0.006 (0.1513)
  Calcium; Week 24; n=123 | 0.007 (0.1440)
  Cholesterol; Week 4; n=132 | -0.034 (0.7416)
  Cholesterol; Week 8; n=126 | -0.062 (0.8776)
  Cholesterol; Week12; n=126 | -0.180 (0.9450)
  Cholesterol; Week 16; n=126 | -0.281 (0.8570)
  Cholesterol; Week 20; n=125 | -0.277 (0.8482)
  Cholesterol; Week 24; n=121 | -0.253 (0.8340)
  Chloride; Week 4; n=131 | 0.48 (7.594)
  Chloride; Week 8; n=127 | 1.02 (3.858)
  Chloride; Week12; n=127 | 1.51 (3.409)
  Chloride; Week 16; n=126 | 1.01 (3.995)
  Chloride; Week 20; n=124 | 1.40 (3.715)
  Chloride; Week 24; n=123 | 1.32 (4.758)
  Glucose; Week 4; n=130 | -0.343 (1.7140)
  Glucose; Week 8; n=126 | -0.222 (1.7264)
  Glucose; Week12; n=126 | -0.263 (1.7351)
  Glucose; Week 16; n=126 | -0.218 (1.9083)
  Glucose; Week 20; n=124 | -0.133 (1.5598)
  Glucose; Week 24; n=121 | -0.246 (1.4132)
  Potassium; Week 4; n=132 | -0.208 (0.4190)
  Potassium; Week 8; n=127 | -0.169 (0.4690)
  Potassium; Week12; n=127 | -0.188 (0.4834)
  Potassium; Week 16; n=126 | -0.223 (0.5053)
  Potassium; Week 20; n=124 | -0.147 (0.5728)
  Potassium; Week 24; n=123 | -0.168 (0.4538)
  Magnesium; Week 4; n=124 | 0.007 (0.0860)
  Magnesium; Week 8; n=121 | 0.008 (0.0900)
  Magnesium; Week12; n=119 | 0.008 (0.1032)
  Magnesium; Week 16; n=118 | 0.002 (0.0986)
  Magnesium; Week 20; n=116 | -0.005 (0.0988)
  Magnesium; Week 24; n=113 | 0.007 (0.0990)
  Sodium; Week 4; n=132 | 0.43 (3.196)
  Sodium; Week 8; n=127 | 0.53 (3.270)
  Sodium; Week12; n=127 | 1.01 (3.048)
  Sodium; Week 16; n=126 | 0.54 (3.361)
  Sodium; Week 20; n=124 | 0.84 (3.050)
  Sodium; Week 24; n=123 | 0.58 (4.485)
  Inorganic Phosphorus; Week 4; n=129 | -0.064 (0.2729)
  Inorganic Phosphorus; Week 8; n=124 | -0.085 (0.3164)
  Inorganic Phosphorus; Week12; n=124 | -0.058 (0.4237)
  Inorganic Phosphorus; Week 16; n=123 | -0.075 (0.3298)
  Inorganic Phosphorus; Week 20; n=121 | -0.091 (0.2792)
  Inorganic Phosphorus; Week 24; n=120 | -0.037 (0.5258)
  Triglycerides; Week 4; n=131 | -0.116 (0.6109)
  Triglycerides; Week 8; n=127 | -0.079 (0.5917)
  Triglycerides; Week12; n=126 | -0.119 (0.7142)
  Triglycerides; Week 16; n=126 | -0.124 (0.8533)
  Triglycerides; Week 20; n=124 | -0.211 (0.6071)
  Triglycerides; Week 24; n=122 | -0.222 (0.6796)
  Urea/BUN; Week 4; n=133 | -0.438 (1.5434)
  Urea/BUN; Week 8; n=127 | -0.527 (1.9777)
  Urea/BUN; Week12; n=127 | -0.542 (1.8160)
  Urea/BUN; Week 16; n=126 | -0.655 (1.8838)
  Urea/BUN; Week 20; n=125 | -0.821 (1.8408)
  Urea/BUN; Week 24; n=123 | -0.635 (1.9606)

25. Secondary Outcome: Number of Participants With Urinalysis Data at Baseline and Week 24
Description: Urine samples were collected for urinalysis at Baseline and Week 24. The Number of participants with urinalysis to negative and positives (trace, +, ++ and +++) data at Baseline and Week 24 are summarized for urine bilirubin (UBIL), urine glucose (UGLU), urine ketones (UKET), urine nitrite (UNIT), urine protein (UM) and urine urobilinogen (UUBIL) were performed with dipstick method. Other urinalysis parameters included urine pH (UpH), urine specific gravity (USG). The Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline and Week 24
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 134
Participants
  UBIL; Baseline; negative | 125
  UBIL; Baseline; positive | 7
  UBIL; Week24; negative | 102
  UBIL; Week 24; positive | 8
  UGLU; Baseline; negative | 132
  UGLU; Baseline; positive | 0
  UGLU; Week24; negative | 109
  UGLU; Week 24; positive | 1
  UKET; Baseline; negative | 126
  UKET; Baseline; positive | 6
  UKET; Week24; negative | 101
  UKET; Week 24; positive | 9
  UNIT; Baseline; negative | 129
  UNIT; Baseline; positive | 3
  UNIT; Week24; negative | 108
  UNIT; Week 24; positive | 2
  UM; Baseline; negative | 87
  UM; Baseline; positive | 45
  UM; Week24; negative | 73
  UM; Week 24; positive | 37
  UUBIL; Baseline; negative | 109
  UUBIL; Baseline; positive | 23
  UUBIL; Week24; negative | 95
  UUBIL; Week 24; positive | 15

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of administration of the study drug (up to Week 24)
Description: SAEs and non-serious AEs were reported for members of the safety population, comprised of all participants who had received at least one dose of study medication.
Arm/Group | Ambrisentan
Serious Adverse Events (participants affected / at risk) | 11/134
Other Adverse Events (participants affected / at risk) | 59/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=134)
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Sudden cardiac death (General disorders) | 2
Oedema peripheral (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cystitis glandularis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=134)
Oedema peripheral (General disorders) | 15
Flushing (Vascular disorders) | 11
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 7
Headache (Nervous system disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 6
Dizziness (Nervous system disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Blood glucose increased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.